CLINICAL TRIAL: NCT04188054
Title: Reducing Knee Compression Loading When Sleeping Supine (on the Back): Benefits in Patients With Knee Osteoarthritis
Brief Title: Reducing Knee Compression When Sleeping in Those With Knee OA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bradford (Other)
Responsible Party: Principal Investigator, John G Buckley, Principal Investigator, University of Bradford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 241876; 18/YH/0057 (Other: Research Ethics Committee)
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will be asked to change the position they lie on their bed when sleeping; that is, to re-position themselves when lying on their back so that their feet (and ankles) hang over the end of the mattress.
  Interventions: Behavioral: Change in sleeping position
- Control (Placebo Comparator): Will be asked to make no change in the way they normally lie on their mattress when sleeping
  Interventions: Behavioral: No change in sleeping position

INTERVENTIONS:
Behavioral: Change in sleeping position — The new sleeping position requires you to re-position yourself in your bed when lying on your back so that your feet (and ankles) hang over the end of the mattress, i.e. off the end of the bed.
  Arms: Intervention
Behavioral: No change in sleeping position — No change to your normal sleeping position
  Arms: Control

SUMMARY:
To determine whether a change in sleeping position so as to prevent the knee being 'pushed' into full extension when lying supine provides pain relief and/or symptom improvement in individuals with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Only those who normally sleep lying on their back will be recruited. Participants will be recruited into two groups: Group 1, 'intervention'; Group 2, 'control'. Participants in group 1 will be asked to change the position they lie on their bed when sleeping; that is, to re-position themselves when lying on their back so that their feet (and ankles) hang over the end of the mattress. Participants in group 2 will be asked to make no change in the way they normally lie on their mattress when sleeping.

Participants will be asked to complete a questionnaire, asking them about the pain and/or discomfort they are currently experiencing, and their current level of physical functioning. The questionnaire used will be the Knee Injury and Osteoarthritis Outcome Score (KOOS) which has been widely used to assess intervention outcomes in individuals with knee OA. They will be asked to complete this questionnaire three times over a 4-month period; for Group 1 this will be before (x2) and after (x1) changing to the new sleeping position (i.e. day of consent, 1 month later on day of change, and 3 months after change); for Group 2 this will be matching the intervals in the intervention group. The primary outcome measure will be the KOOS Pain score, which will be compared pre and post- changing to the new sleeping position.

ELIGIBILITY:
Inclusion Criteria:

* presence of mild, moderate or severe tibiofemoral-OA (radiologically determined in either or both knees)
* regularly (routinely) spend periods lying on their back when sleeping.

Exclusion Criteria:

* those with: rheumatoid arthritis
* chronic cardiopulmonary problems
* lower-limb joint(or joint surface) replacement and/or previous knee surgery within previous 12 months
* unable to lie supine in bed (medical or practical reason)
* diagnosed with inflammatory arthropathy
* peripheral neuropathy or other sensory problems
* steroid injection in the knee within previous 3 months
* under 18 years of age
* unable to give consent due to lack of mental capacity
* currently involved in any research study related to knee OA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
change in KOOS Knee Pain | baseline and 3 months (post intervention)
  Knee injury and Osteoarthritis Outcome Scores (KOOS) - sub-scale Pain, from 0 (worst) to 100 (best)

SECONDARY OUTCOMES:
change in KOOS Knee (other sub-scales) | baseline and 3 months (post intervention)
  Knee injury and Osteoarthritis Outcome Scores (KOOS) subscales: Symptoms; Activities-of-Daily-Living; Quality-of-Life, from 0 (worst) to 100 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Idle Medical Centre, Bradford, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No